CLINICAL TRIAL: NCT03640130
Title: Factors Limiting Peripheral Reading
Brief Title: Peripheral Reading
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Daniel R. Coates, Assistant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001096
Record Dates: First submitted 2018-08-19; First posted 2018-08-21 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Central Visual Impairment
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Each participant will participate in several blocks (randomized order), to evaluate performance with and without behavioral gaze-contingent text enhancements.
  Interventions: Behavioral: Gaze-contingent text enhancement

INTERVENTIONS:
Behavioral: Gaze-contingent text enhancement — In different testing blocks, the efficacy of the different enhancements will be evaluated, such as inverting the text in a gaze-contingent inverted "spotlight."

SUMMARY:
The purpose of this study is to evaluate reading performance in the visual periphery by simulating central vision loss using a computer-controlled gaze-contingent display with an eye tracker. Participants will read a page of text at a comfortable rate. Several manipulations hypothesized to improve reading will be tested, such as an inverted-text "spotlight" of a single word that follows the participant's gaze.

DETAILED DESCRIPTION:
Participants will view paragraphs of multiple sentences of text with their central vision blocked computationally with a "simulated scotoma." Participants will be free to move their eyes around the page of text at a comfortable rate. The three outcomes described elsewhere will be evaluated.

In different blocks, text will contain one or more of several dynamic assistive manipulations that are hypothesized to enhance reading: 1) inverting the text at a given position, with instructions for the participant to attend to that location, which simulates a "surrogate fovea" of a patient with central vision loss. 2) horizontally expanding text to alleviate within-word crowding. 3) highlighting the next word with a visible indicator to encourage proper eye movements.

ELIGIBILITY:
Inclusion Criteria:

* Normal vision
* English language

Exclusion Criteria:

* Less than 20/20 vision in either eye
* Abnormalities which affect vision (amblyopia, keratoconus, etc.)
* Ortho-K lenses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Reading speed | From enrollment to completion of testing (<2 weeks)
  Average time/word it takes to read a paragraph of text.
Reading accuracy | From enrollment to completion of testing (<2 weeks)
  Ability to correctly answer comprehension questions or orally read words
Efficiency of eye movement | From enrollment to completion of testing (<2 weeks)
  Ability to move the eyes systematically from word to word

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
To conform with open science directives, will likely post the de-identified behavioral data on a public server.